CLINICAL TRIAL: NCT03679468
Title: Improving Cognition in People With Progressive Multiple Sclerosis: A Multi-Arm, Randomized, Blinded, Sham-Controlled Trial of Cognitive Rehabilitation and Aerobic Exercise.
Brief Title: Improving Cognition in People With Progressive Multiple Sclerosis Using Aerobic Exercise and Cognitive Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Florence (Other); Fondazione Italiana Sclerosi Multipla (Other); University College, London (Other); Kessler Foundation (Other); University of Alabama at Birmingham (Other); University of Southern Denmark (Other); Hasselt University (Other); University of Plymouth (Other); Universita degli Studi di Genova (Other); Unity Health Toronto (Other); Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Dr. Anthony Feinstein, Professor, department of psychiatry, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 232-2018
Record Dates: First submitted 2018-08-23; First posted 2018-09-20 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis, Primary Progressive; Cognitive Impairment
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Cognitive Dysfunction | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Intervention Model Description: We propose undertaking a randomized, blinded, sham controlled clinical trial investigating the effectiveness of CR and exercise, either singly or in combination, in treating cognitive dysfunction in people with progressive MS. Subjects will be randomly assigned to one of four groups: CR plus exercise; CR plus passive exercise; passive CR plus exercise and passive CR plus passive exercise. Subjects will receive one of these four treatments for 12 weeks, twice a week. One in three subjects will undergo structural and functional MRI to investigate how the brain responds to the two interventions.
Who Masked: Participant, Investigator
Masking Description: In order to prevent bias in our research results, we will employ a double-blind study design in which the examiner nor the research participant will know which group membership they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Rehab & Sham Exercise (Sham Comparator): Cognitive Rehabilitation by computer based brain tasks, and Sham exercises focusing primary on balance and stretching. Sessions will take place twice a week for 12 weeks.
  Interventions: Other: Cognitive Rehabilitation; Other: Sham Exercise
- Sham Cognitive Rehab & Sham Exercise (Sham Comparator): Sham cognitive Rehabilitation will consist of basic internet searches and learning to use a computer, and sham exercises focusing primary on balance and stretching. Sessions will take place twice a week for 12 weeks.
  Interventions: Other: Sham Exercise; Other: Sham Cognitive Rehabilitation
- Sham Cognitive rehab & Aerobic Exercise (Sham Comparator): Sham cognitive rehabilitation will consist of basic internet searches and learning to use a computer, and aerobic exercises will focus primarily on improving cardio-respiratory fitness using a recumbent bike. Sessions will take place twice a week for 12 weeks.
  Interventions: Other: Sham Cognitive Rehabilitation; Other: Aerobic Exercise
- Cognitive Rehab & Aerobic Exercise (Active Comparator): Cognitive Rehabilitation by computer based brain tasks and aerobic exercises will focus primarily on improving cardio-respiratory fitness using a recumbent bike. Sessions will take place twice a week for 12 weeks.
  Interventions: Other: Cognitive Rehabilitation; Other: Aerobic Exercise

INTERVENTIONS:
Other: Cognitive Rehabilitation — RehaCom software
  Information processing speed and attention modules
  Arms: Cognitive Rehab & Aerobic Exercise; Cognitive Rehab & Sham Exercise
Other: Sham Exercise — Sets of balance and stretching exercises
  Arms: Cognitive Rehab & Sham Exercise; Sham Cognitive Rehab & Sham Exercise
Other: Sham Cognitive Rehabilitation — Kompozer software
  24 session module consisting of basic internet searches
  Arms: Sham Cognitive Rehab & Sham Exercise; Sham Cognitive rehab & Aerobic Exercise
Other: Aerobic Exercise — Recumbent NuStep Bike
  Aerobic cycling
  Arms: Cognitive Rehab & Aerobic Exercise; Sham Cognitive rehab & Aerobic Exercise

SUMMARY:
Given that up to 70% of people with secondary progressive MS are cognitively impaired, the search for effective treatments is considered a priority by people living with the disease. This proposal will address the effectiveness of cognitive rehabilitation (CR) and exercise, either alone, or in combination in this regard. A team of MS researchers has been assembled from the USA, Canada, the United Kingdom, Italy, Denmark, Germany and Belgium for this. A total of 360 people with progressive MS will make up the sample. Brain MRIs will be undertaken in a third of the sample before and after the 12 weeks of treatment to document the functional changes that are expected to occur with symptom improvement.

DETAILED DESCRIPTION:
Aim: The broad aim of this proposal is to evaluate a multidisciplinary and multi-modal approach to rehabilitation in people with progressive MS. Cognitive rehabilitation and aerobic exercise will be evaluated individually and in combinations to address cognitive dysfunction as the primary outcome variable.

Over 20 years have passed since the introduction of the first disease modifying treatment, interferon beta-1betaseron (b), for multiple sclerosis (MS).Since then 13 treatments have been approved and made it onto the market. All are for relapsing-remitting disease (RRMS), apart from mitoxantrone which is limited to progressive disease with relapses, Interferon-beta-1b, which is for secondary progressive disease (SPMS), but does not delay disability progression and Ocrelizumab for primary progressive MS only. Thus, for a sizeable proportion of people with MS there is no therapeutic option to slow progression. This raises the question, how are patients with primary and secondary progressive MS (PPMS and SPMS) to be helped? While research is underway to find a medication that holds promise of halting further deterioration in a disease that has already entered a progressive stage, patients and their clinicians are left with basically symptomatic treatments.

Hypothesis: The investigators hypothesize that CR and aerobic exercise are effective treatments for cognitive impairment (processing speed deficits) in people with progressive MS. In particular a combination of these two treatment given twice weekly over 12 weeks is more effective than each individual treatment given alone or as sham. The investigators further hypothesize that improvements in processing speed will be matched on functional MRI (fMRI) by enhanced neural activity in networks associated with information processing speed.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed diagnosis of progressive Multiple Sclerosis
* Visual Acuity of 20/70
* Language comprehension, to ensure subjects have the ability to understand instructions

Exclusion Criteria:

* Wheelchair dependent (EDSS > 7.0)
* History of central nervous system disease other than progressive MS
* Steroids use within the past 3 months
* Regular aerobic training (eg. bi-cycling, running, swimming or rowing)
* Unwilling to travel to study sites for rehabilitation 2 times a week for 3 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline cognitive Information processing speed at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  The Symbol Digit Modalities Test (SDMT) will be used to measure cognitive information processing speed
  The SDMT is a simple matching task that requires the participant to refer to a reference key, in order to correctly match a geometric symbol with the corresponding number. Participant will be under a 90 second time constraint to quickly and correctly match each pair.
  Test will be administered at index assessment, 12 weeks following cognitive rehab/ aerobic exercise, and at 6 months to examine cognitive retention

SECONDARY OUTCOMES:
Change from baseline cognitive verbal memory at 12 weeks and 6 months | Baseline, 12 weeks, & 6 month
  The California Verbal Learning Test (CVLT) will be used to measure verbal memory
  The CVLT test begins with the examiner reading a list of 16 words, participants are then instructed to report as many of the words as they can remember. After recall is recorded, the entire list is read again, altogether, there are five learning trials.
  Test will be administered at index assessment, 12 weeks following cognitive rehab/ aerobic exercise, and at 6 months to examine cognitive retention
Change from baseline cognitive visual memory at 12 weeks and 6 months | Baseline, 12 weeks, & 6 month
  The Brief Visuo-Spatial Memory Test (BVMT) will be used to measure visual memory
  Participants are presented with six abstract designs for 10 seconds, the display is then removed from view and participant are instructed to draw the designs from memory via pencil on paper. Each design is scored from 0 to 2 points representing accuracy and location. There are three learning trials.
  Test will be administered at index assessment, 12 weeks following cognitive rehab/ aerobic exercise, and at 6 months to examine cognitive retention
Change from baseline anxiety & depression, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  The following self report scale will be used to measure anxiety and depression:
  The Hospital Anxiety and Depression Scale (HADS) - The HADS is comprised of seven questions for anxiety and seven questions for depression, each reply has a likert scale ranging from 0-3.
  Total score will indicate:
  0-7 = normal 8-10 = borderline abnormal 11-21 = abnormal
Change from baseline depression, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  The following self report scale will be used to measure depression:
  Beck Depression Inventory-revised (BDI-II) - The BDI-II questionnaire is comprised of 21 questions, participant will circle a reply that closely matches their answer, each reply has a likert scale that ranges from 0-3.
  Total score indicate the following:
  1-10 = these ups and downs are considered normal 11-16 = Mild mood disturbance 17-20 = Borderline clinical depression 21-30 = Moderate depression 31-40 = Severe depression over 40 = Extreme depression
Change from baseline fatigue, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  Self report scale:
  The Modified Fatigue Impact Scale (MFIS), will evaluate the participants fatigue.
  The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.
Change from baseline perceived deficits, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  Self report scale:
  The Perceived Deficits Questionnaire (PDQ), will evaluate the participants subjective cognitive difficulties.
  The total score for the PDQ is the sum of the scores for the 20 items. Individual subscale scores for attention/concentration, retrospective memory, prospective memory, and planning/organization will be generated by calculating the sum of specific sets of items.
Change from baseline subjective impact of walking, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  Self report scale:
  The Multiple Sclerosis Walking Scale (MSWS-12), will evaluate the participants subjective impact of walking.
  The MSWS-12 consist of 12 questions, each question ranges from 0-5. A high total score indicates greater impact on walking than lower scores.
Change from baseline impact of Multiple Sclerosis, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  Self report scale:
  Multiple Sclerosis Impact Scale (MSIS-29-V2) - will evaluate the participants impact of Multiple Sclerosis.
  The MSIS-29 is a 29 item scale measuring the physical (20 item) and psychological (9 item) impact of Multiple scleroses.
Change from baseline quality of life, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  Self report scale:
  European Quality of Life-5 Dimensions (EQ5D-5) - will be used to evaluate the participants quality of life.
  The EQ5D-5 comprises of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
  The EQ5D-5 also records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine".
Change from baseline global function, at 12 weeks and 6 months | Baseline, 12 weeks, and 6 month
  Self report scale:
  The Functional Assessment of Multiple Sclerosis (FAMS), will be used to asses the participants global function.
  The FAMS consist of 59 items, and domains that consist of questions on: mobility, symptoms, emotional well-being, general contentment, thinking/fatigue, family/social well-being, and additional concerns.
  FAMS total score range = 0 -176. Higher scores indicate better quality of life.

OTHER OUTCOMES:
Change from baseline brain activity at 12 weeks and 6 months | Baseline, 12 weeks, 6 months
  The participant will perform a modified Go no Go task while in the MRI. Changes in brain activity will indicate superiority of one of the four study groups.
  Go no Go task:
  Participants are required to either respond (i.e., pressing designated key) or withhold a response (not pressing designated key) depending on whether a go stimulus or a no-go stimulus is presented
  MRI Go no Go task will be administered at index assessment, 12 weeks following cognitive rehab/ aerobic exercise, and at 6 months to examine brain activity and anatomical changes

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Feinstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Science Center, Toronto, Ontario, Canada

REFERENCES:
- [Result] Feinstein A, Amato MP, Brichetto G, Chataway J, Chiaravalloti N, Dalgas U, DeLuca J, Feys P, Filippi M, Freeman J, Meza C, Inglese M, Motl RW, Rocca MA, Sandroff BM, Salter A, Cutter G; CogEx Research Team. Study protocol: improving cognition in people with progressive multiple sclerosis: a multi-arm, randomized, blinded, sham-controlled trial of cognitive rehabilitation and aerobic exercise (COGEx). BMC Neurol. 2020 May 22;20(1):204. doi: 10.1186/s12883-020-01772-7. PMID 32443981
- [Result] Feinstein A, Amato MP, Brichetto G, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell R, Feys P, Filippi M, Freeman J, Inglese M, Meza C, Motl RW, Rocca MA, Sandroff BM, Salter A; CogEx Research Team. Cognitive rehabilitation and aerobic exercise for cognitive impairment in people with progressive multiple sclerosis (CogEx): a randomised, blinded, sham-controlled trial. Lancet Neurol. 2023 Oct;22(10):912-924. doi: 10.1016/S1474-4422(23)00280-6. PMID 37739574
- [Result] Feinstein A, Amato MP, Brichetto G, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell R, Feys P, Filippi M, Freeman J, Inglese M, Meza C, Motl R, Rocca MA, Sandroff BM, Salter A; CogEx Research Team. The impact of the COVID-19 pandemic on an international rehabilitation study in MS: the CogEx experience. J Neurol. 2022 Apr;269(4):1758-1763. doi: 10.1007/s00415-021-10881-3. Epub 2021 Nov 5. PMID 34741240
- [Result] Feinstein A, Amato MP, Brichetto G, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell R, Feys P, Filippi M, Freeman J, Inglese M, Meza C, Motl RW, Rocca MA, Sandroff BM, Salter A; CogEx Research Team. The late onset of emotional distress in people with progressive multiple sclerosis during the Covid-19 pandemic: longitudinal findings from the CogEx study. J Neurol. 2022 Dec;269(12):6202-6210. doi: 10.1007/s00415-022-11295-5. Epub 2022 Aug 8. PMID 35939096
- [Result] Feinstein A. The CogEx trial - Cognitive rehabilitation and aerobic exercise for cognitive impairment in people with progressive multiple sclerosis: A randomised, blinded, sham-controlled trial. Mult Scler. 2023 Nov;29(13):1523-1525. doi: 10.1177/13524585231210178. Epub 2023 Nov 2. No abstract available. PMID 37916484
- [Result] Sandroff BM, Motl RW, Amato MP, Brichetto G, Chataway J, Chiaravalloti ND, Cutter GR, Dalgas U, DeLuca J, Farrell R, Feys P, Filippi M, Freeman J, Inglese M, Meza C, Rocca MA, Salter A, Feinstein A. Cardiorespiratory fitness and free-living physical activity are not associated with cognition in persons with progressive multiple sclerosis: Baseline analyses from the CogEx study. Mult Scler. 2022 Jun;28(7):1091-1100. doi: 10.1177/13524585211048397. Epub 2021 Oct 1. PMID 34595972
- [Result] Chiaravalloti ND, Amato MP, Brichetto G, Chataway J, Dalgas U, DeLuca J, Meza C, Moore NB, Feys P, Filippi M, Freeman J, Inglese M, Motl R, Rocca MA, Sandroff BM, Salter A, Cutter G, Feinstein A; CogEx Research Team. The emotional impact of the COVID-19 pandemic on individuals with progressive multiple sclerosis. J Neurol. 2021 May;268(5):1598-1607. doi: 10.1007/s00415-020-10160-7. Epub 2020 Aug 19. PMID 32813051
- [Result] Veldkamp R, D'hooge M, Sandroff BM, DeLuca J, Kos D, Salter A, Feinstein A, Amato MP, Brichetto G, Chataway J, Farrell R, Chiaravalloti ND, Dalgas U, Filippi M, Freeman J, Motl RW, Meza C, Inglese M, Rocca MA, Cutter G, Feys P; CogEx Research Team. Profiling cognitive-motor interference in a large sample of persons with progressive multiple sclerosis and impaired processing speed: results from the CogEx study. J Neurol. 2023 Jun;270(6):3120-3128. doi: 10.1007/s00415-023-11636-y. Epub 2023 Mar 7. PMID 36881147
- [Result] Romano F, Motl RW, Valsasina P, Amato MP, Brichetto G, Bruschi N, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell R, Feys P, Freeman J, Inglese M, Meza C, Salter A, Sandroff BM, Feinstein A, Rocca MA, Filippi M; CogEx Research Team. Abnormal thalamic functional connectivity correlates with cardiorespiratory fitness and physical activity in progressive multiple sclerosis. J Neurol. 2023 Jun;270(6):3213-3224. doi: 10.1007/s00415-023-11664-8. Epub 2023 Mar 18. PMID 36933030
- [Result] Preziosa P, Rocca MA, Pagani E, Valsasina P, Amato MP, Brichetto G, Bruschi N, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell R, Feys P, Freeman J, Inglese M, Meani A, Meza C, Motl RW, Salter A, Sandroff BM, Feinstein A, Filippi M; the CogEx Research Team. Structural and functional magnetic resonance imaging correlates of fatigue and dual-task performance in progressive multiple sclerosis. J Neurol. 2023 Mar;270(3):1543-1563. doi: 10.1007/s00415-022-11486-0. Epub 2022 Nov 27. PMID 36436069
- [Derived] Romano F, Rocca MA, Pagani E, Amato MP, Brichetto G, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell R, Feys P, Freeman J, Inglese M, Cipriano E, Meza C, Motl RW, Salter A, Sandroff BM, Feinstein A, Filippi M; CogEx Research Team. Effects of cognitive rehabilitation and exercise on brain structure in progressive multiple sclerosis: results from the CogEx trial. J Neurol. 2025 Sep 23;272(10):645. doi: 10.1007/s00415-025-13382-9. PMID 40986118
- [Derived] Rocca MA, Valsasina P, Romano F, Tedone N, Amato MP, Brichetto G, Boccia VD, Chataway J, Chiaravalloti ND, Cutter G, Dalgas U, DeLuca J, Farrell RA, Feys P, Freeman J, Inglese M, Meza C, Motl RW, Salter A, Sandroff BM, Feinstein A, Filippi M; Cogex Research Team. Cognitive rehabilitation effects on grey matter volume and Go-NoGo activity in progressive multiple sclerosis: results from the CogEx trial. J Neurol Neurosurg Psychiatry. 2024 Nov 18;95(12):1139-1149. doi: 10.1136/jnnp-2024-333460. PMID 38754979
- [Derived] Ramari C, D'hooge M, Dalgas U, Feinstein A, Amato MP, Brichetto G, Chataway J, Chiaravalloti ND, Cutter GR, DeLuca J, Farrell R, Filippi M, Freeman J, Inglese M, Meza C, Motl RW, Rocca MA, Sandroff BM, Salter A, Kos D, Feys P. Prevalence and Associated Clinical Characteristics of Walking-Related Motor, Cognitive, and Fatigability in Progressive Multiple Sclerosis: Baseline Results From the CogEx Study. Neurorehabil Neural Repair. 2024 May;38(5):327-338. doi: 10.1177/15459683241236161. Epub 2024 Mar 1. PMID 38426484